CLINICAL TRIAL: NCT01763437
Title: Intralesional Tetracycline Injection in the Treatment of Chalazia
Acronym: TET
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TET2013
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Chalazia; Chalazion
Keywords: Chalazia; Chalazion; Meibomian gland dysfunction; Rosacea; Ocular rosacea
MeSH Terms: conditions — Chalazion; Meibomian Gland Dysfunction; Rosacea | interventions — Tetracycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): 30 patients will be randomized to observation alone. These patients will return 4 weeks (+/- 2 weeks) after their initial visit for lesion measurement and photographs.
- Tetracycline (Experimental): 30 patients will be randomized to treatment with an intralesional injection of 0.05 mL of 2% tetracycline solution. These subjects will return 4 weeks (+/- 2 weeks) after treatment for lesion measurement and photographs.
  Interventions: Drug: Tetracycline

INTERVENTIONS:
Drug: Tetracycline — Chalazia randomized to the treatment arm will be injected with 0.05 mL of 2% tetracycline solution.
  Arms: Tetracycline

SUMMARY:
The investigators propose a study to investigate the role of tetracycline injection into chalazia versus observation alone. The investigators hypothesize tetracycline injection will result in a significant decrease in lesion size when compared to observation alone.

DETAILED DESCRIPTION:
Intralesional Tetracycline Injection in the Treatment of Chalazia

Authors: Bryan R. Costin, M.D. and Julian D. Perry, M.D.

Purpose: To investigate the therapeutic role of intralesional tetracycline injection when compared to observation alone in the treatment of chalazia.

Introduction:

The tetracycline family includes tetracycline, doxycycline, and minocycline and this group of compounds has a surprising number of properties including but not limited to antibiotic, anti-malarial, anti-inflammatory, and antioxidant. Recent applications include uses both in sclerotherapy in a wide variety of conditions from ganglions cysts to lymphangiomas to ovarian cysts as well as in the reduction of hypertrophic scarring in rabbit models.1,2,3,4 In 2009, there were approximately 130 ongoing clinical trials studying this class of drugs in an astounding variety of conditions from gingivitis to Alzheimer disease to brain cancer.5

Chalazia are lipogranulomatous inflammatory lesions of the eyelid and are one of the most common eyelid lesions and an extremely frequent presenting complaint to the ophthalmologist. Chalazia often represent significant morbidity for the patients suffering from these lesions because they are often recurrent, can be refractory to treatment, and are disfiguring. Consequently, chalazia can also be a challenge to the ophthalmologist. Oral tetracyclines have been shown to be effective in the treatment of ocular rosacea and meibomian gland dysfunction (MGD), which are conditions commonly seen in association with chalazia. The anti-inflammatory effect of the tetracyclines is thought to be beneficial in rosacea and these drugs have been shown to alter the fatty acid composition of the lipid layer of the tear film perhaps explaining their efficacy in MGD.6

Chalazia eventually resolve without intervention, but the process can take many months and patients are frequently dissatisfied with observation as a treatment modality. Often patients choose incision and drainage (I&D) of the lesion and this method is often successful. Another treatment shown to be effective in chalazion treatment is the injection of corticosteroid directly into the lesion, hence providing a depot anti-inflammatory effect.7 However, unlike corticosteroids, the tetracyclines would offer antibiotic, sclerosant, and lipid tear film augmentation, in addition to their anti-inflammatory effect. Further, tetracyclines are FDA approved for the treatment of acne8, which is defined as inflammation of pilosebaceous units9, and chalazia are defined as inflammation of sebaceous glands10. With these multiple roles in mind, we propose injection of tetracycline into chalazia to investigate its use as a multipurpose depot.

Methods:

After IRB approval, chalazia patients who wish to participate will be enrolled after the risks, benefits, alternatives, and personnel have been explained to them and informed consent has been obtained. A total of 80 subjects will be randomized to one of two groups: 40 subjects to observation alone and 40 subjects to treatment with an intralesional injection of 0.05 mL 2% tetracycline solution. Subjects will be excluded from the study if they are less than 18 years of age, are pregnant, have chalazia of less than 1 week duration, have known allergies to tetracycline or its derivatives, or are currently taking oral tetracyclines or have taken them in the past 3 months. Men, post-menopausal women, and women who have undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy will not be tested for pregnancy. Pregnancy testing (urine or serum) will be performed on women of childbearing age before enrollment and the results checked prior to the administration of treatment.

For patients with multiple lesions, either on the same or opposite eyelids, only the most symptomatic lesion will be enrolled in the study. Eyelid margin disease and ocular rosacea will be documented at the time of enrollment. Subjects will then be examined at 4 weeks (+/- 2 weeks) post-procedure follow-up visits where data regarding lesion size, including color photography, lesion regression or recurrence, and a complete ophthalmic examination will be recorded. If subjects fail to follow up at any of these visits, telephone interviews will be conducted.

At the time of enrollment, the subject's date of birth, sex, race/ethnicity, and last menstrual period will be determined as well as a gynecological history to determine need for pregnancy testing. Data collection sheets will be used to record information. Also, previous therapies including topical medications and previous surgeries will be reviewed. A millimeter ruler will be used at the time of enrollment to determine the size of the lesion. Lesion photographs will also be taken so that the independent chalazion photograph reviewer will be able to grade degrees of improvement after treatment in a masked fashion.

When the procedure is performed, a variable pain scale will be used by the patient to document their level of discomfort during the injection. At the return post procedure visit, the lesion will be re-measured, the patient will be asked to grade the level of improvement and a follow up photograph will be taken for use by the masked grader. All data collection sheets and consents will be stored at the Cleveland Clinic in a secure location. All other study data will be electronic and stored only on the secure Cleveland Clinic server or Cleveland Clinic issued encrypted devices such as thumb drives and laptops. The occurrence of any minor adverse or unexpected events will be reported to the principal investigator. Any sentinel events will be reported to the IRB immediately.

A decrease in lesion size by two-thirds of greater as determined by either the clinician or the masked photograph reviewer in either group will be considered improvement and if seen in lesions injected with tetracycline it will constitute treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Not pregnant
* Chalazia of greater than 1 week duration
* Not allergic to tetracycline or its derivatives
* Not currently taking tetracycline or not taking them in the past 3 months

Exclusion Criteria:

* Age less than 18 years old
* Pregnancy
* Chalazia of less than 1 week duration
* Allergies to tetracycline or its derivatives
* Currently taking tetracyclines or have taken them in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Lesion size | 4 weeks
  The size of the lesion will be measured as well as photographed. Photographs will be reviewed by a masked chalazion photograph reviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Julian D Perry, M.D., Principal Investigator — Cleveland Clinic Cole Eye Institute
Locations (1):
- Cleveland Clinic Cole Eye Institute, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ashindoitiang JA. Preliminary report of the effectiveness of tetracycline sclerotherapy in treatment of ganglion. Plast Surg Int. 2012;2012:624209. doi: 10.1155/2012/624209. Epub 2012 Mar 26. PMID 22570781
- [Background] Chaudry G, Burrows PE, Padua HM, Dillon BJ, Fishman SJ, Alomari AI. Sclerotherapy of abdominal lymphatic malformations with doxycycline. J Vasc Interv Radiol. 2011 Oct;22(10):1431-5. doi: 10.1016/j.jvir.2011.06.021. Epub 2011 Aug 6. PMID 21821431
- [Background] Kars B, Buyukbayrak EE, Karsidag AY, Pirimoglu M, Unal O, Turan C. Comparison of success rates of 'transvaginal aspiration and tetracycline sclerotherapy' versus 'only aspiration' in the management of non-neoplastic ovarian cysts. J Obstet Gynaecol Res. 2012 Jan;38(1):65-9. doi: 10.1111/j.1447-0756.2011.01627.x. Epub 2011 Aug 10. PMID 21827579
- [Background] Henry SL, Concannon MJ, Kaplan PA, Diaz-Arias AA. The inhibitory effect of minocycline on hypertrophic scarring. Plast Reconstr Surg. 2007 Jul;120(1):80-88. doi: 10.1097/01.prs.0000263325.73400.f8. PMID 17572548
- [Background] Griffin MO, Fricovsky E, Ceballos G, Villarreal F. Tetracyclines: a pleitropic family of compounds with promising therapeutic properties. Review of the literature. Am J Physiol Cell Physiol. 2010 Sep;299(3):C539-48. doi: 10.1152/ajpcell.00047.2010. Epub 2010 Jun 30. PMID 20592239
- [Background] Souchier M, Joffre C, Gregoire S, Bretillon L, Muselier A, Acar N, Beynat J, Bron A, D'Athis P, Creuzot-Garcher C. Changes in meibomian fatty acids and clinical signs in patients with meibomian gland dysfunction after minocycline treatment. Br J Ophthalmol. 2008 Jun;92(6):819-22. doi: 10.1136/bjo.2007.133900. Epub 2008 May 29. PMID 18511542
- [Background] Ben Simon GJ, Huang L, Nakra T, Schwarcz RM, McCann JD, Goldberg RA. Intralesional triamcinolone acetonide injection for primary and recurrent chalazia: is it really effective? Ophthalmology. 2005 May;112(5):913-7. doi: 10.1016/j.ophtha.2004.11.037. PMID 15878075
- [Result] Lacy CF, Armstrong LL, Goldman, MP, Lance LL. Lexi-Comp's Drug Information Handbook. 13th ed. 2005. 1447.
- [Result] Wolff K, Johnson RA, et al. Fitzpatrick's Color Atlas & Synopsis of Clinical Dermatology. 5th ed. McGraw-Hill. 2005.
- [Result] Macquire JI, Murchinson AP, et al. Wills Eye Institute 5-minute Ophthalmology Consult. Lippencott Williams & Wilkins.